CLINICAL TRIAL: NCT00060567
Title: Phase I Dose-Finding Study of E7070 in Combination With Irinotecan
Brief Title: Dose-Finding Study of E7070 in Combination With Irinotecan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7070-A001-106
Record Dates: First submitted 2003-05-07; First posted 2003-05-09 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2013-06

CONDITIONS: Cancer
Keywords: E7070; Irinotecan; hydrochloride; gastrointestinal; cancer
MeSH Terms: conditions — Neoplasms | interventions — N-(3-chloro-7-indolyl)-1,4-benzenedisulphonamide; Irinotecan

ARMS (3):
- 1 (Other): Active combination of E7070 and irinotecan.
  Interventions: Drug: E7070 + irinotecan combination
- 2 (Other): Active combination of E7070 and irinotecan.
  Interventions: Drug: Irinotecan + E7070 combination
- 3 (Other): Active combination of E7070 and irinotecan.
  Interventions: Drug: Irinotecan + E7070 combination

INTERVENTIONS:
Drug: E7070 + irinotecan combination — Escalating doses starting from 125 mg/m2 irinotecan plus 250 mg/m2 E7070 combination.
  Arms: 1
Drug: Irinotecan + E7070 combination — Escalating doses starting from 100 mg/m2 irinotecan plus 400 mg/m2 E7070 combination.
  Arms: 2
Drug: Irinotecan + E7070 combination — Escalating doses starting from 100 mg/m2 irinotecan plus 400 mg/m2 E7070 combination.
  Arms: 3

SUMMARY:
E7070 and irinotecan will be administered to patients with GI tract, pancreatic or lung tumors on Days 1 and 8 of a 21-day cycle, or Days 1 and 15 of a 28-day cycle according to one of two E7070 dose escalation schemes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically or cytologically confirmed refractory small cell lung carcinoma or relapsed pancreatic cancer.
2. Patients should not have received more than two previous regimens of chemotherapy (prior epidermal growth factor directed therapy antiangiogenic therapy, or capecitabine do not constitute a previous regimen),
3. Patients must be aged greater than or equal to 18 years,
4. Patients must be ambulatory and have a Karnofsky performance status greater than or equal to 70%,
5. Patients must have a life expectancy of greater than or equal to 3 months,
6. Patients must meet the following screening hematologic values:

   * Hemoglobin greater than or equal to 10g /dL
   * Absolute Neutrophil Count greater than or equal to 1.5 x 10^9/L
   * Platelets greater than or equal to 100 x 109/L,
7. Patients must meet the following screening values for liver function:

   * Serum bilirubin less than or equal to 1.5 x upper limits of normal (ULN)
   * ALAT and ASAT less than or equal to 2.5 x ULN (unless related to liver metastases, in which case less than or equal to 5 x ULN),
8. Patients must have serum creatinine less than or equal to 1.5 x ULN,
9. Patients must be willing and able to comply with the study protocol for the duration of the study, and
10. Patients must give written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.

Exclusion Criteria:

1. Patients who have received chemotherapy or radiation therapy (except palliative) or who have had major surgery within four weeks of treatment start,
2. Patients who have received chemotherapy without recovering from chemotherapy related toxicity (defined as grade 1 or less) at study entry,
3. Patients who have received palliative radiation therapy without recovering from radiation associated toxicity at study entry,
4. Patients with a history of hypersensitivity to irinotecan,
5. Patients who experienced greater than or equal to Grade 3 toxicity during previous therapy with irinotecan,
6. Women who are pregnant or breastfeeding. Women of childbearing potential with either a positive pregnancy test at screening or no pregnancy test. Women of childbearing potential unless (1) surgically sterile or (2) using adequate measures of contraception in the opinion of the Investigator (postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential),
7. Fertile men who are not willing to use contraception or fertile men with a female partner who is not willing to use contraception,
8. Any history of uncontrolled seizures; CNS disorders; or psychological, familial, sociological or geographical conditions, judged by the Investigator to be clinically significant, and/or potentially capable of precluding informed consent or adversely affecting compliance with the study protocol and follow-up schedule,
9. Patients must not have untreated brain metastases (Patients who have been treated for CNS metastases must be asymptomatic and radiologically stable for 4 weeks prior to entry),
10. Patients with a history of conjugated hyperbilirubinemia,
11. Patients with clinically significant cardiac or cardiovascular impairment,
12. Patients with severe uncontrolled intercurrent infections,
13. Patients with organ allografts,
14. Patients who are receiving investigational drug treatment, immunotherapy, or biologic therapy. Treatment must have been completed four weeks prior to entry into the study and patients must have recovered from any associated toxicity.
15. Patients with a history of hypersensitivity to sulfonamides,
16. Patients with surgically resectable metastatic disease,
17. Patients who are known to be positive for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), Hepatitis C antibody, or human immunodeficiency virus,
18. Patients with significant disease, in the Investigator's opinion, that would exclude the patient from the study,
19. Patients who are legally incapacitated,
20. Patients who have a repeated demonstration of QTc greater than 470 ms (Bazett's correction),
21. Patients with tumor, including metastasis, that is surgically resectable,
22. Patients with clinical symptoms from brain metastasis,
23. Patients taking steroids for the treatment of brain metastases, or
24. Patients with leptomeningeal metastasis,
25. Patients who have a history of additional risk factors for torsades de pointes (e.g., heart failure) or family history of Long QT Syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2003-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To determine the Maximum tolerated dose of E7070 in combination with irinotecan in patients with GI tract, pancreatic or lung tumors. | 1st arm: D1, D8, Q3WK; 2nd arm: D1, D8, Q3WK; 3rd arm: D1, D15, Q4WK

SECONDARY OUTCOMES:
Safety, E7070 activity and Pharmacokinetics | 1st arm: D1, D8, Q3WK; 2nd arm: D1, D8, Q3WK; 3rd arm: D1, D15, Q4WK

CONTACTS AND LOCATIONS:
Overall Officials: Eisai Medical Services, Study Director — Eisai Inc.
Locations (1):
- Boston, Massachusetts, United States